CLINICAL TRIAL: NCT05396612
Title: Role of the Immune Environment in Response to Therapy in Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Jennifer Zhang, Assistant Professor of Surgery, Abramson Cancer Center at Penn Medicine
Other Study IDs: UPCC 19121; 850338 (Other: University of Pennsylvania)
Record Dates: First submitted 2022-05-05; First posted 2022-05-31 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; ER Positive Breast Cancer; HER2-negative Breast Cancer; TNBC - Triple-Negative Breast Cancer
Keywords: Immune microenvironment
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue from breast tumors removed as standard of care treatment for breast cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Collection of personal health information from women treated at the University of Pennsylvania under an approved HIPAA waiver. — Collection of personal health information from women treated at the University of Pennsylvania under an approved HIPAA waiver.

SUMMARY:
This is an observational case-control study of tissues collected from women with ER+HER2- breast cancers. The immune environments of these cancers will be compared to triple negative and HER2+ breast cancers. No randomization or changes to standard of care treatment will occur as part of the study.

ELIGIBILITY:
Inclusion criteria:

Women 18 years of age or older with non-metastatic breast cancer undergoing surgical resection in the University of Pennsylvania Health System.

Exclusion criteria:

Males Children Pregnant individuals

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women 18 years of age or older undergoing surgery for breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Collecting, processing and archiving breast cancer tumor tissues | Through study completion, average of 2 years
  This study will collect and analyze tumor samples from women diagnosed with primary breast cancer. The investigators will dissociate fresh tumor samples and analyze single cell suspensions by flow cytometry. Percentage of dendritic cell and T cell subsets and dendritic cell and T cell activation markers will be compared between breast cancer subtypes (HR+HER2-, HER2+, triple negative). Percentage of dendritic cell and T cell subsets and dendritic cell and T cell activation markers will be compared between HR+HER2- untreated breast cancers compared to HR+HER2- chemotherapy treated breast cancers.

SECONDARY OUTCOMES:
Associating breast cancer dendritic cell infiltrate with outcome | 5 years
  We will perform studies to associate dendritic cell infiltration and activation markers with patient outcome, including disease free survival, distant disease free survival, and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Zhang, MD, Principal Investigator — Abramson Cancer Center
Locations (1):
- Abramson Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.